CLINICAL TRIAL: NCT05819437
Title: Effectiveness of a 3-week Balneotherapy Program With Mineral Water of Saint Jean d'Angely in Knee Osteoarthritis: A Superiority, Randomised, Controlled Study Versus Standard of Care Alone
Brief Title: Knee Osteoarthritis and Balneotherapy
Acronym: ANGELLO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CEN Biotech (Industry)
Collaborators: COMPAGNIE EUROPEENNE DES BAINS (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: C1650
Record Dates: First submitted 2023-04-06; First posted 2023-04-19 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Knee Osteoarthritis
Keywords: Balneotherapy, Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Intervention Model Description: Randomized controlled Trial, monocentric
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CONTROL (No Intervention): Standard of care for knee osteoarthritis
- BALNEOTHERAPY PROGRAM (Experimental): 3-week balneotherapy program with Mineral Water of Saint Jean d'Angely in addition to standard of care for knee osteoarthritis
  Interventions: Other: Balneotherapy program

INTERVENTIONS:
Other: Balneotherapy program — Whirlpool bath, bath with immersion showers, poultice application and underwater massage.
  The baths were performed in an individual tub in ten-minute sessions. The temperature was set specifically for each patient, on average from 34 to 38°C. These were baths with jets and air diffusion.
  The mud was applied as a poultice to the 2 knees and if necessary (duration of application: 10 minutes).
  The massages were carried out by qualified physiotherapists under an affusion ramp of thermal water at 38°C for 10 minutes.
  The water used is a mixed sulphated Natural Mineral Water, collected by drilling the "capuchins" at a depth of 975 m. The temperature of the water at the outlet of the borehole is 41.8°C and is lowered to 35°C.
  Arms: BALNEOTHERAPY PROGRAM

SUMMARY:
The goal of this clinical trial is to assess the efficacy of a 18-day balneotherapy program in the rheumatology indication in patients presented with knee osteoarthritis. The main questions of the study aims to answer are how balneotherapy improves functional incapacity and the disorders (pain, joint stiffness) induced by osteoarthritis of the knee, and thus improves patients' quality of life.

Participants are randomly assigned in control or treatment (spa) groups. All receive standard of care for knee osteoarthritis throughout the study. Balneotherapy program consists of 18-days of spa treatment with Mineral Water of Saint Jean d'Angely. Functional incapacity, disorders and quality of life induced were measured at baseline and then 6 months later.

Variation from baseline were compared in control and treatment groups to assess the efficacy of the balneotherapy program.

ELIGIBILITY:
Inclusion Criteria:

* Knee osteoarthritis with Kellgren and Lawrence stage 2 to 4 evidenced by a knee X-ray examination in the past 3 years);
* 100-normalized score of the WOMAC physical function subscale of 30 or greater;
* Available for balneotherapy program and the 6-month study follow-up;
* Signed inform consent;
* with health insurance affiliation.

Exclusion Criteria:

* Presented with balneotherapy contra-indication;
* Having had spa treatment in the past 6 months or intra-articular corticosteroid injection within the previous 90 days or hyaluronic acid infiltration within the previous 6 months;
* Presented with chronic pain other than osteoarthritis, with scheduled surgery related to knee osteoarthritis;
* regulatory reason (guardianship or already enrolled in a clinical trial).

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2020-08-26 (Actual); Primary Completion 2021-07-03 (Actual); Study Completion 2022-09-20 (Actual)

PRIMARY OUTCOMES:
Variation from baseline in physical function subscale of the WOMAC at 6 months | Baseline (D1) and final (6 months)
  Physical function subscale of the Western Ontario and McMaster Universities Arthritis Index (WOMAC) is a self-administered questionnaire that consists in 17 items: (17 items): using stairs, rising from sitting, standing, bending, walking, getting in / out of a car, shopping, putting on / taking off socks, rising from bed, lying in bed, getting in / out of bath, sitting, getting on / off toilet, heavy domestic duties, light domestic duties. The 100-normalized subscale score ranges from 0 (none) to 100 (worse functional limitations).

SECONDARY OUTCOMES:
Variation from baseline in physical function subscale of the WOMAC at 3 months | Baseline (D1) and final (3 months)
  Physical function subscale of the Western Ontario and McMaster Universities Arthritis Index (WOMAC) is a self-administered questionnaire that consists in 17 items: (17 items): using stairs, rising from sitting, standing, bending, walking, getting in / out of a car, shopping, putting on / taking off socks, rising from bed, lying in bed, getting in / out of bath, sitting, getting on / off toilet, heavy domestic duties, light domestic duties. The 100-normalized subscale score ranges from 0 (none) to 100 (worse functional limitations).
Variation from baseline in pain subscale of the WOMAC at 3 months | Baseline (D1) and final (3 months)
  Pain subscale of the WOMAC is a self-administered questionnaire that consists in 5 items: during walking, using stairs, in bed, sitting or lying, and standing upright. The 100-normalized subscale score ranges from 0 (none) to 100 (worse pain limitations).
Variation from baseline in pain subscale of the WOMAC at 6 months | Baseline (D1) and final (6 months)
  Pain subscale of the WOMAC is a self-administered questionnaire that consists in 5 items: during walking, using stairs, in bed, sitting or lying, and standing upright. The 100-normalized subscale score ranges from 0 (none) to 100 (worse pain limitations).
Variation from baseline in stiffness subscale of the WOMAC at 3 months | Baseline (D1) and final (3 months)
  Stiffness subscale of the WOMAC is a self-administered questionnaire that consists in 2 items: during walking, using stairs, in bed, sitting or lying, and standing upright. The 100-normalized subscale score ranges from 0 (none) to 100 (worse stiffness limitations).
Variation from baseline in stiffness subscale of the WOMAC at 6 months | Baseline (D1) and final (6 months)
  Stiffness subscale of the WOMAC is a self-administered questionnaire that consists in 2 items: during walking, using stairs, in bed, sitting or lying, and standing upright. The 100-normalized subscale score ranges from 0 (none) to 100 (worse stiffness limitations).
Variation from baseline in WOMAC total score at 3 months | Baseline (D1) and final (3 months)
  The scores for each subscale are summed up to calculate the total WOMAC score. The 100-normalized score ranges from 0 (none) to 100 (worse limitations).
Variation from baseline in WOMAC total score at 6 months | Baseline (D1) and final (6 months)
  The scores for each subscale are summed up to calculate the total WOMAC score. The 100-normalized score ranges from 0 (none) to 100 (worse limitations).
Variation from baseline in pain-induced knee osteoarthritis intensity at 3 months | Baseline (D1) and final (3 months)
  Pain intensity is measured using a 0 (no pain)-100 (Worse pain) Visual Analogic Scale (VAS).
Variation from baseline in pain-induced knee osteoarthritis intensity at 6 months | Baseline (D1) and final (6 months)
  Pain intensity is measured using a 0 (no pain)-100 (Worse pain) Visual Analogic Scale (VAS).
Number of participants achieving minimal clinically important improvement (MCII) at 3 months | 3 months
  MCII is defined as 19.9 mm or greater on the VAS pain scale and/or 9.1 points or greater on the WOMAC physical function subscale normalized to a 0-100 score, and no knee surgery
Number of participants achieving minimal clinically important improvement (MCII) at 6 months | 6 months
  MCII is defined as 19.9 mm or greater on the VAS pain scale and/or 9.1 points or greater on the WOMAC physical function subscale normalized to a 0-100 score, and no knee surgery
Number of participants presented with acceptable symptom state (ASS) at 3 months | 3 months
  ASS is defined as VAS pain 32 mm or less or WOMAC function subscale normalized to a 0-100 score of 31 points or less.
Number of participants presented with acceptable symptom state (ASS) at 6 months | 6 months
  ASS is defined as VAS pain 32 mm or less or WOMAC function subscale normalized to a 0-100 score of 31 points or less.
Changes in participants quality of life at 3 months | 3 months
  Quality of life is measured using EUROQOL (EQ-5D-3L) questionnaire.The EQ-5D-3L descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results into a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
Changes in participants quality of life at 6 months | 6 months
  Quality of life is measured using EUROQOL (EQ-5D-3L) questionnaire.The EQ-5D-3L descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results into a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
Frequency of adverse events throughout the study | From inclusion to the final visit at 6 months
  Adverse events are described using MedDRA and each event frequency is calculated.
Participants' opinion with their symptoms related to knee osteoarthritis at 6 months | 6 months
  Opinion is measured using a 5-point Likert scale

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud TERRILLON-SEYTRE, Study Director — CEN
Locations (1):
- CEN, Dijon, France

IPD SHARING:
Plan to Share IPD: No